CLINICAL TRIAL: NCT00335465
Title: Pilot Study for the Evaluation of the Effects of Insulin Treatment on Myocardial Function, Perfusion, and Glucose Metabolism in Patients With Primary Left Ventricular Dysfunction and Type 2 Diabetes.
Brief Title: Lantus Effect on Myocardial Glucose Metabolism in T2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4053; EUDRACT # : 2004-002729-34
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Insulin glargine — once a daily, sc injection, 100IU/ml

SUMMARY:
The primary objective of the present study is to assess changes of myocardial glucose uptake (MGU) during clamp studies using positron emission tomography (PET) scanning in patients with type 2 diabetes and idiopathic left ventricular dysfunction (LVD).

The secondary objectives of the study are: assessment of changes of myocardial microcirculation at rest and during adenosine stimulation using PET; assessment of changes in myocardial structure and function evaluated by magnetic resonance imaging (MRI); assessment of glycaemic control by measurement of HbA1c, fasting blood glucose and insulin levels; assessment of safety (adverse event profile, laboratory data).

ELIGIBILITY:
Inclusion Criteria:

* LV systolic dysfunction (2D-Echo LVEF < 50%) with or without LV dilation (2D-Echo LV EDD > 56 mm) or left ventricular end-diastolic diameter (LVEDD) >55mm with or without LV dysfunction
* angiographically normal coronary arteries (< 50% vessel narrowing);
* newly diagnosed type 2 diabetes;
* previously diagnosed: OAD treated type 2 diabetic patients able to take part in the study after a one-month wash-out period and insulin treated type 2 diabetic patients able to take part in the study after one week wash-out period.

Exclusion Criteria:

* evidence of congenital or valvular cardiac diseases, hypertrophic cardiomyopathy, overt heart failure (NYHA class III-IV);
* moderate to severe hypertension (diastolic aortic pressure > 100 mmHg);
* hypotension (systolic aortic pressure < 100 mmHg);
* nephropathy (serum creatinine > 3 mg/dL);
* other systemic and/or infective diseases;
* severe dyslipidemia;
* peripheral vasculopathy;
* necessity of vasoactive medical treatment in the last 48 hours;
* atrial fibrillation;
* Refusal or impossibility to give written informed consent;
* patients diagnosed with type 1 insulin dependent diabetes;
* clinically relevant cardiovascular, hepatic, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult;
* patients with medical history positive for cerebrovascular accidents, including Transient Ischaemic Attack (TIA);
* women who are lactating, pregnant, or planning to become pregnant during the study;
* history of hypersensitivity to the investigational products or to drugs with similar chemical structures;
* likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol;
* treatment with any investigational product in the last 30 days or 5 half-lives (whichever is longer) before study entry;
* current use of investigational agents or participation in any other investigational studies during study period;
* history of drug or alcohol abuse;
* impaired hepatic function, as shown by Alamine AminoTransferase (ALT) > 2,5 times the upper limit of the normal laboratory range;
* mental condition making the subject unable to understand the nature, scope, and possible consequences of the study;
* patients unable to understand dosing directions;
* subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study procedures;
* receipt of an experimental drug or use of an experimental device within the 30 days prior to study entry;
* previous enrollment in the present study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
effect of insulin treatment on myocardial function, perfusion and glucose metabolism. | assessed before and after treatment
adverse events | throughout the study

SECONDARY OUTCOMES:
changes of myocardial structure and left ventricular systolic and diastolic function | at baseline and at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Georges Paizis, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Milan, Italy

REFERENCES:
- [Derived] Masi S, Lautamaki R, Guiducci L, Di Cecco P, Porciello C, Pardini S, Morales MA, Chubuchny V, Salvadori PA, Emdin M, Sironi AM, Knuuti J, Neglia D, Nuutila P, Ferrannini E, Iozzo P. Similar patterns of myocardial metabolism and perfusion in patients with type 2 diabetes and heart disease of ischaemic and non-ischaemic origin. Diabetologia. 2012 Sep;55(9):2494-500. doi: 10.1007/s00125-012-2631-0. Epub 2012 Jul 1. PMID 22752026